CLINICAL TRIAL: NCT04838522
Title: A Breast Milk Study in Lactating Women Who Have Been Prescribed Therapeutic Doses of MOTEGRITY® or RESOTRAN® (Prucalopride) for Chronic Idiopathic Constipation to Evaluate Prucalopride Concentrations in Breast Milk, and to Collect Incidental Safety Data From the Nursing Infants
Brief Title: A Study of Prucalopride in Breastfeeding Women With Constipation
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: UC San Diego Human Milk Research Biorepository (Unknown)
Responsible Party: Sponsor
Other Study IDs: TAK-555-4006; EUPAS40105 (Other: EUPAS Register Number)
Record Dates: First submitted 2021-03-25; First posted 2021-04-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Chronic Idiopathic Constipation (CIC)
Keywords: Prucalopride; Motegrity; Pharmacokinetics; Lactation; Breastfeeding; Milk-only study; Infant growth and development; Infant neurodevelopment; Infant outcomes
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Study Participants: Participants with chronic idiopathic constipation who are treated with prucalopride oral tablets which was initiated prior to enrollment, and are breastfeeding their infant at the time of enrollment and sample collection will be observed prospectively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
Prucalopride is a medicine used to treat constipation. The main aim of the study is to measure prucalopride concentrations in breast milk. Other aims are to check the growth and development of babies breastfed by their mothers who took prucalopride and to check if the babies had any side effects.

During the study, participants will provide one set of milk samples over 24 hours using an electric breast pump. Breast milk samples will be collected at home and will be shipped to the laboratory.

Also, participants will be asked questions during telephone interviews every 2 months in the first year of their baby's life. They will also be asked to complete growth and development questionnaires about their baby.

ELIGIBILITY:
Inclusion Criteria:

Participants cannot be enrolled before all inclusion criteria are confirmed.

* Female participants with an ability to voluntarily provide verbal followed by written, signed, and dated (personally or via a legally authorized representative) informed consent as applicable to participate in the study.
* Participants greater than or equal to (>=) 18 years of age at the time of consent. This inclusion criterion will only be assessed at the time of enrollment.
* Participants who are currently breastfeeding a singleton infant who is between 10 days and 11 months 0 days, inclusive. Note that participants pumping breast milk and bottle feeding their infant breast milk are allowed to participate.
* Participants who are currently exclusively breastfeeding or breastfeeding with supplemental formula and/or solid food. Infants who are exclusively breastfed and do not yet eat solid food are preferred.
* Participants who are currently treated as prescribed by their physician with MOTEGRITY or RESOTRAN (generic forms of prucalopride not allowed) for functional constipation, including chronic idiopathic constipation (CIC) and irritable bowel syndrome-constipation (IBS-C), for at least 5 consecutive days at the time of taking the first breastmilk sample.
* Participants who agree to the conditions and requirements of the study including the sample collection, interview schedule, completion of developmental questionnaires, and release of medical records.
* Participants with an understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

The participant will be excluded from the study if any of the following exclusion criteria are met:

* Participants who are breastfeeding an infant who: is hospitalized, has a major birth defect, or has a history of a disease that could affect absorption or drug disposition.
* Participants who have used MOTEGRITY or RESOTRAN while breastfeeding for a condition other than functional constipation.
* Participants who are pregnant at the time of enrollment.
* Participants who have started to wean their child from breast milk.
* Participants with a history of any hematological, hepatic, respiratory, cardiovascular, renal, gall bladder removal, or other current or recurrent disease that could affect the action, absorption, or disposition of prucalopride.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female participants from United State (US) and Canada, who are currently being treated with prucalopride for functional constipation and breastfeeding a single infant between the ages of 10 days and 11 months 0 days. Infants will be followed for up to 12 months 30 days of age.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose- Normalized Area Under the Milk Concentration-time Curve of Prucalopride (AUC [milk, norm]) | Pre-dose, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 1
  AUC [milk, norm] will be derived from a series of 7 timed, full expression breast milk samples collected from a single breast using an electric breast pump over a 24-hour period of milk collection after a dose following at least 5 consecutive daily doses. AUC [milk, norm] will be normalized to 2-milligrams (mg) daily maternal dose.
Dose- Normalized Average Concentration of Prucalopride in Milk (C [ave, milk, norm]) | Pre-dose, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 1
  C [ave, milk, norm] will be derived from a series of 7 timed, full expression breast milk samples collected from a single breast using an electric breast pump over a 24-hour period of milk collection after a dose following at least 5 consecutive daily doses. C [ave, milk, norm] will be normalized to 2-mg daily maternal dose.
Time Interval Over Which the AUC [milk, norm] Measured (T) | Pre-dose, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 1
  Time interval over which the AUC [milk, norm] is measured (T) will be reported.
Dose-normalized Daily Infant Dosage (DID [norm]) | Pre-dose, 1, 2, 4, 8, 12, and 24 hours post-dose
  DID [norm] will be the estimated daily infant dose received by the infant through breastfeeding. DID [norm] will be normalized to 2-mg daily maternal dose.
Percentage of Maternal Dose or Relative Infant Dose (RID [%]) | Up to 24 hours post-dose
  RID [%]will be calculated as DID [norm] divided by (2 mg/day/maternal body weight (kg)) then multiplied by 100.

SECONDARY OUTCOMES:
Number of Infants With Adverse Events (AEs) Based on Maternal Report | Up to 1 year of age
  Number of infants with AEs while being breastfed by a mother who is taking prucalopride will be obtained by maternal report (by phone).
Change in Length During the First Year of Life in Infant's | At 6 and 12 months of age
  Growth changes in length in centimeters every 2 months during the first year of life in infant's breastfed by mothers taking prucalopride will be obtained by maternal report (by phone), and medical records abstraction.
Change in Weight During the First Year of Life in Infant's | At 6 and 12 months of age
  Growth changes in weight in grams every 2 months during the first year of life in infant's breastfed by mothers taking prucalopride will be obtained by maternal report (by phone), and medical records abstraction.
Change in Head Circumference During the First Year of Infant's Life | At 6 and 12 months of age
  Change in head circumference at 6 and 12 months will be reported.
Infant's Neurodevelopmental Performance Based on Ages and Stages Questionnaire-3 (ASQ-3) | Up to 1 year of age
  Infant's neurodevelopmental progress at 12 months will be assessed by the ASQ-3 which will be completed by the mother. The ASQ-3 is a developmental screening instrument with 5 domains: (i) personal-social, (ii) gross motor, (iii) fine motor, (iv) problem solving, and (v) communication. All domains will be evaluated both continuously and categorically, with 3 categories: normal, borderline, abnormal. Abnormal scores of clinical concern are defined by test-based, standardized scoring criteria reported in the ASQ-3 User's Guide; these represent scores that are <2.0 SDs below the mean for each category. Borderline scores are scores that fall between 2.0 and 1.5 SDs below the mean. Each domain has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. ASQ-3 average = average score of 5 aspects.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda; Study Director, Study Director — UC San Diego Human Milk Research Biorepository
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/607462db688ad8001f42fb8e
- Available data/document: Breast Milk At the Dawn of New Discoveries — https://betterbeginnings.org/what-we-do/research/breast-milk/